CLINICAL TRIAL: NCT05493644
Title: A Study About the Selection of Time for Retreatment of Helicobacter Pylori After Eradication Failure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Professor, Director of gastroenterology department of Qilu hospital, Shandong University
Other Study IDs: 2022-SDU-QILU-G808
Record Dates: First submitted 2022-08-08; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- group A: Within 3 months of treatment failure in the course of Helicobacter pylori infection,Patients will receive esomeprazole (Nexium) 40mg po bid, bismuth potassium citrate(Lizhudele) 220mg po bid, amoxicillin1000mg po bid and tetracycline 500 mg po qid (or tetracycline 500 mg po tid) for 14d.
  Interventions: Other: Remedial treatment within 3 months
- group B: Within 3 to 6 months of treatment failure in the course of Helicobacter pylori infection,Patients will receive esomeprazole (Nexium) 40mg po bid, bismuth potassium citrate(Lizhudele) 220mg po bid, amoxicillin1000mg po bid and tetracycline 500 mg po qid (or tetracycline 500 mg po tid) for 14d.
  Interventions: Other: Remedial treatment within 3 to 6 months
- group C: Within 6 to 12 months of treatment failure in the course of Helicobacter pylori infection,Patients will receive esomeprazole (Nexium) 40mg po bid, bismuth potassium citrate(Lizhudele) 220mg po bid, amoxicillin1000mg po bid and tetracycline 500 mg po qid (or tetracycline 500 mg po tid) for 14d.
  Interventions: Other: Remedial treatment within 6 to 12 months
- group D: After 12 months of treatment failure in the course of Helicobacter pylori infection,Patients will receive esomeprazole (Nexium) 40mg po bid, bismuth potassium citrate(Lizhudele) 220mg po bid, amoxicillin1000mg po bid and tetracycline 500 mg po qid (or tetracycline 500 mg po tid) for 14d.
  Interventions: Other: Remedial treatment after 12 months

INTERVENTIONS:
Other: Remedial treatment within 3 months — Remedial therapy was performed within 3 months
  Groups: group A
Other: Remedial treatment within 3 to 6 months — Remedial therapy was performed within 3 to 6 months
  Groups: group B
Other: Remedial treatment within 6 to 12 months — Remedial therapy was performed within 6 to 12 months
  Groups: group C
Other: Remedial treatment after 12 months — Remedial therapy was performed after 12 months
  Groups: group D

SUMMARY:
The patients who accepted the quadruple eradication program of the helicobacter pylori but failed to eradicate helicobacter pylori will be assessed the most suitable re-eradication time of helicobacter pylori.

DETAILED DESCRIPTION:
Helicobacter pylori (HP) infection is a common global infectious disease, which is an important cause of chronic gastritis, peptic ulcer and gastric cancer. At present, due to the non-standard Helicobacter pylori eradication program in clinical work, poor patient compliance and other reasons, the phenomenon of HP eradication treatment failure is more and more common. However, there is still no conclusion on the most appropriate time for remedial treatment inpatients with Hp eradication failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 with H. pylori infection.
* Patients with previous Helicobacter pylori eradication.

Exclusion Criteria:

* Patients treated with H2-receptor antagonist, PPI, bismuth and antibioticsin the previous 4 weeks.
* Patients with gastrectomy, acute GI bleeding and advanced gastric cancer.
* Patients with known or suspected allergy to study medications.
* Currently pregnant or lactating.
* Inability to provide informed consent and other situations that couldinterfere with the examination or therapeutic protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-70 with previous Helicobacter pylori eradication failure.
Sampling Method: Non-Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The most suitable re-eradication time | 12 months
  The most suitable re-eradication time#The unit is month# will be assessed by paired comparison method .

SECONDARY OUTCOMES:
Eradication rates in three groups | 12 months
  Both intention to treat(ITT) and per-protocol(PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in three groups